CLINICAL TRIAL: NCT03054506
Title: A Randomized, Single Center, Double-blind, Parallel-group, Placebo-controlled Study Assessing the Effect of CSP01 on Chronic Idiopathic Constipation and Irritable Bowel Syndrome With Constipation
Brief Title: The Effect of CSP01 on Chronic Idiopathic Constipation and Irritable Bowel Syndrome With Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Gelesis, Inc. (Industry)
Responsible Party: Principal Investigator, Kyle Staller, MD, MPH, Kyle Staller, MD, MPH, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P001751
Record Dates: First submitted 2017-02-07; First posted 2017-02-15 (Actual); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Constipation; Chronic Idiopathic Constipation; Irritable Bowel Syndrome With Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- CSP01 (Experimental): Subjects in the experimental group will receive CSP01, a non-systemic, orally administered hydrogel capsule, twice a day. CSP01 capsules are taken prior to a meal with water, after which the small particles within the capsules hydrate and expand in the stomach and small intestine. By acting as a bulking agent and possibly reducing colonic transit time through increase of colonic water content, CSP01 may contribute to constipation relief.
  Interventions: Device: CSP01
- Carboxymethylcellulose (CMC) (Active Comparator): Subjects in the active control group will receive orally administered 3 capsules of carboxymethylcellulose (CMC) capsules twice a day.
  Interventions: Device: Carboxymethylcellulose (CMC)
- Placebo (Placebo Comparator): Matching placebo consists of an inert mixture supplied by Gelesis Inc. in identical-appearing capsules.Subjects in the placebo group will be administered 3 capsules of placebo twice a day.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: CSP01 — Subjects will take three capsules in the morning before breakfast, and three capsules at night before dinner each day for three weeks.
  Arms: CSP01
Device: Carboxymethylcellulose (CMC) — Subjects will take three capsules in the morning before breakfast, and three capsules at night before dinner each day for three weeks.
  Arms: Carboxymethylcellulose (CMC)
Device: Placebo — Subjects will take three capsules in the morning before breakfast, and three capsules at night before dinner each day for three weeks.
  Arms: Placebo

SUMMARY:
Constipation is a common gastrointestinal motility disorder that is often chronic, negatively affects patients' daily lives. Constipation occurs when bowel movements become difficult or less frequent.This study is being done to study the effectiveness of the hydrogel capsule, CSP01, compared to the active control (carboxymethylcellulose) and placebo (non-medicine sugar pill), to relieve constipation among subjects with chronic idiopathic constipation (CIC) or with irritable bowel syndrome with constipation (IBS-C).

ELIGIBILITY:
Inclusion Criteria:

1. Age 22-70 years old
2. BMI >18.5 and <35 kg/m2
3. Rome III criteria for functional constipation or IBS-C
4. Continued IBS-C or CIC throughout Run-in period
5. Compliant with reporting during Run-in (confirm the presence of constipation during the 7-day Run-in baseline period; patients are required to report an average of <3 continuous spontaneous bowel movements [CSBMs] and ≤6 spontaneous bowel movements [SBMs] per week via the interactive web response system).
6. Ability to follow verbal and written instructions
7. Ability to record daily bowel habits, including frequency, stool consistency (BSFS), straining (EoPS), completeness of evacuation, and Patient Reported Outcomes (PROs) (abdominal discomfort, severity of constipation, bloating, overall relief)
8. Informed consent form signed by the subjects

Exclusion Criteria:

1. History of loose stools
2. History of irritable bowel syndrome with diarrhea (IBS-D) or mixed irritable bowel syndrome (IBS-M)
3. Non-compliance with reporting during Run-in
4. Patients reporting laxative, enema, and/or suppository usage for >2 days or any usage of a prohibited medication during the Run-in period
5. Patients reporting watery stools for any SBM (Type 7 on the Bristol Stool Form Scale [BSFS]) or loose (mushy) stools for >1 SBM (Type 6 on the BSFS) in the absence of laxatives during Run-in
6. GI motility obstruction or GI tract structural abnormality
7. Current use of prescribed or illicit opioids
8. History of pelvic floor dysfunction
9. Need for manual maneuvers in order to achieve a BM
10. History of GI lumen surgery at any time or other GI or abdominal operations within 60 days prior to entry into the study
11. History of high-dose stimulative or cathartic laxative abuse as judged by investigator team
12. Neurological disorders, metabolic disorders, or other significant disease that would impair their ability to participate in the study
13. Cardiovascular disease, diabetes, cancer, Crohn's disease, ulcerative colitis
14. BMI of <18.5 or >35 kg/m2
15. Pregnancy (or positive serum or urine pregnancy test(s) in females of childbearing potential) or lactation
16. Absence of contraception in females of childbearing potential
17. History of allergic reaction to carboxymethylcellulose, citric acid, sodium stearyl fumarate, raw cane sugar, gelatin, or titanium dioxide
18. Administration of investigational products within 1 month prior to Screening Visit
19. Exclusion of colonic inertia with symptoms of < 1 BM per 2 weeks
20. Subjects anticipating surgical intervention during the study
21. Known history of diabetes (type 1 or 2)
22. History of eating disorders including binge eating (except mild binge eater)
23. Supine SBP > 160 mm Hg and/or supine DBP > 95 mm Hg (mean of two consecutive readings)
24. Angina, coronary bypass, or myocardial infarction within 6 months prior to Screening Visit
25. History of swallowing disorders
26. Esophageal anatomic abnormalities (e.g., webs, diverticuli, rings)
27. History of gastric bypass or any other gastric surgery
28. History of small bowel resection (except if related to appendectomy)
29. History of gastric or duodenal ulcer
30. History of gastroparesis
31. History of abdominal radiation treatment
32. History of pancreatitis
33. History of intestinal stricture (e.g., Crohn's disease)
34. History of intestinal obstruction or subjects at high risk of intestinal obstruction including suspected small bowel adhesions
35. History of malabsorption
36. History of sucrose intolerance
37. History of hepatitis B or C
38. History of human immunodeficiency virus
39. History of cancer within the past 5 years (except adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer)
40. Any other clinically significant disease interfering with the assessments of Gelesis100, according to the Investigator (e.g., disease requiring corrective treatment, potentially leading to study discontinuation)
41. HbA1c > 8.5% (> 69 mmol/mol)
42. Positive test for drugs in the urine
43. Any relevant biochemical abnormality interfering with the assessments of Gelesis100, according to the Investigator
44. Antidiabetic medications within 1 month prior to Screening Visit (except stable dose of metformin, ≤ 1500 mg/day, for at least 1 month in subjects with type 2 diabetes)
45. Medications requiring mandatory administration with meal at lunch or dinner
46. Anticipated requirement for use of prohibited concomitant medications
47. Implanted or externally worn medical device such as, but not limited to, a pacemaker, infusion pump, or insulin pump

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Staller, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 patients signed the consent form and thus were considered enrolled. 4 failed screening 48 passed screening
  5 withdrew before run-in
  1 lost to follow-up 42 started run-in
  2 failed run-in 40 randomized
  1 withdrew due to AE 39 completed study
  1 patient's follow-up CTT data irretrievable (technical malfunction) 38 complete CTTs
Period: Overall Study
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Started | 20 | 11 | 9
Completed | 19 | 11 | 9
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo | Total
Number analyzed (Participants) | 20 | 11 | 9 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 9 | 8 | 32
  >=65 years | 5 | 2 | 1 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 7 | 35
  Male | 1 | 2 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 20 | 9 | 9 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 2 | 1 | 0 | 3
  White | 16 | 8 | 8 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 11 | 9 | 40
Diagnosis: CIC, IBS-C [Count of Participants; unit: Participants]
  Chronic Idiopathic Constipation | 14 | 9 | 4 | 27
  Irritable Bowel Syndrome with Constipation | 6 | 2 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Colonic Transit Time (CTT)
Description: Colonic Transit Time is the amount of time (in minutes) that the SmartPill capsule spent in the large intestine before expulsion. We measured the difference between CTT pre-treatment and post-treatment and calculated the mean difference for each treatment group. Negative values equal a reduction in CTT.
Time Frame: Up to 1 week; measured once during the run-in-period and again during third week of the treatment period
Population: All participants who completed the study. (39 participants) Note: One participant who received placebo had pre-treatment CTT data, but post-treatment CTT data was irretrievable due to technical malfunction. This subject's pre-treatment CTT data is included in analysis, but no post-treatment CTT data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
minutes | -727 (1277) | -15 (2226) | 366 (1714)

2. Secondary Outcome: Complete Spontaneous Bowel Movement (CSBM) Frequency Rate
Description: Average number of Complete Spontaneous Bowel Movements per day (BMs where participant felt that they emptied their bowels). More CSBMs are interpreted as a better outcome.
Time Frame: 55 days (baseline, treatment, & follow-up)
Population: All participants who completed the study and had both pre and post treatment CSBM measurement
Measure: Mean (Standard Deviation); unit: number of CSBMs per day
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
number of CSBMs per day
  Pre-treatment | 0.2 (0.2) | 0.2 (0.2) | 0.2 (0.3)
  Post-treatment | 0.3 (0.3) | 0.3 (0.2) | 0.3 (0.3)

3. Secondary Outcome: Stool Consistency
Description: Stool consistency for each bowel movement based on the Bristol Stool Scale A descriptive numerical scale from 1 to 7 where lower numbers indicate constipation, numbers toward the middle indicate normal stool consistence, and the highest numbers indicate diarrhea. Therefore middle scores mean a better outcome
  1= hard lumps 2 = lumpy sausage 3 = cracked sausage 4 = smooth sausage 5 = soft lumps 6 = mushy 7 = watery
Time Frame: 55 days (baseline, treatment, & follow-up)
Population: All participants who completed the study and had both pre and post treatment stool consistency ratings.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
score on a scale
  Pre-treatment | 3.62 (0.56) | 3.54 (0.45) | 3.88 (0.65)
  Post-treatment | 3.81 (0.44) | 3.62 (0.59) | 3.59 (0.63)

4. Secondary Outcome: Ease of Passage Rating
Description: Patient assessment of the ease with which bowel movements are passed using a descriptive numerical scale where lower numbers indicate difficult passage of stool, numbers toward the middle indicate more normal passage of stool, and numbers on the highest end indicate abnormally urgent passage of stool. Middle scores indicate a better outcome.
  1. = manual disimpaction needed
  2. = enema needed
  3. = straining needed
  4. = normal
  5. = urgent without pain
  6. = urgent with pain
  7. = incontinent
Time Frame: 55 days (baseline, treatment, & follow-up)
Population: All participants who completed the study and had both pre and post treatment ease of passage ratings
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
score on a scale
  Pre-treatment | 3.62 (0.56) | 3.54 (0.45) | 3.88 (0.65)
  Post-treatment | 3.81 (0.44) | 3.62 (0.59) | 3.59 (0.63)

5. Secondary Outcome: Patient's Assessment of Abdominal Discomfort
Description: Patient's daily assessment of abdominal discomfort using a numerical rating scale of 0 to 10, where 0 = no discomfort at all and 10 = severe discomfort. Higher scores mean a worse outcome.
Time Frame: 55 days (baseline, treatment, & follow-up)
Population: All participants who completed the study and had both pre and post treatment abdominal discomfort ratings
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
score on a scale
  Pre-treatment | 3.91 (1.75) | 3.55 (1.43) | 3.82 (2.23)
  Post-treatment | 3.67 (1.91) | 3.08 (1.41) | 3.58 (2.60)

6. Secondary Outcome: Patient Assessment of Bloating Severity
Description: Patient's daily assessment of bloating severity using a numerical rating scale from 0 to 10 where 0 = no bloating at all and 10 = severe bloating. Higher scores mean a worse outcome.
Time Frame: 55 days (baseline, treatment, & follow-up)
Population: All participants who completed the study and had both pre and post treatment bloating ratings.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
score on a scale
  Pre-treatment | 4.36 (2.20) | 4.43 (1.42) | 4.67 (2.47)
  Post-treatment | 4.17 (2.22) | 3.89 (1.16) | 3.98 (2.80)

7. Secondary Outcome: Patient Assessment of Constipation Severity
Description: Patient's daily assessment of constipation severity using a numerical rating scale from 0 to 10 where 0 = no constipation at all and 10 = severe constipation. Higher numbers mean a worse outcome.
Time Frame: 55 days (baseline, treatment, & follow-up)
Population: All participants who completed the study and had both pre and post treatment constipation severity ratings
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
score on a scale
  Pre-treatment | 4.11 (2.06) | 4.04 (1.34) | 4.15 (2.53)
  Post-treatment | 3.46 (1.77) | 3.29 (1.15) | 3.85 (2.50)

8. Secondary Outcome: Relief Rating
Description: Patient's feeling of overall relief after each bowel movement using a numerical rating scale from 0 to 10 where 0 = no relief and 10 = complete relief. Higher scores mean a better outcome (feeling more relief after a bowel movement).
Time Frame: 55 days (baseline, treatment, & follow-up)
Population: All participants who completed the study and had both pre and post treatment relief ratings
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
score on a scale
  Pre-treatment | 4.27 (1.95) | 4.21 (1.91) | 4.11 (1.78)
  Post-treatment | 5.11 (2.29) | 4.86 (1.99) | 4.38 (1.79)

9. Secondary Outcome: Patient Assessment of Constipation - Symptoms (PAC-SYM)
Description: Patient assessment of constipation symptom severity questionnaire. A validated 12-question questionnaire.
  Numerical scale from 0 to 4 where 0 = absent and 4 = very severe. Possible total score ranges from 0 to 48. Higher total PAC-SYM scores mean a worse outcome.
  PAC-SYM was completed at four time-points (Day -14, Day 0, Day 15, & Day 22). Scores were aggregated based on time period as either pre- (Day -14 & Day 0) or post- (Day 15 & Day 22) treatment start. Values reported are averages based on patient total scores from these time points. Data was specifically analyzed based on patient diagnosis in addition to treatment.
Time Frame: Day -14 to Day 22
Population: All participants who completed the study and had both pre and post treatment PAC-SYM ratings
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
score on a scale
  Pre-treatment (CIC Group): number analyzed (Participants) | 13 | 9 | 4
  Pre-treatment (CIC Group) | 17.62 (6.98) | 17.56 (4.90) | 12.75 (6.85)
  Post-treatment (CIC Group): number analyzed (Participants) | 13 | 9 | 4
  Post-treatment (CIC Group) | 11.77 (7.43) | 9.22 (4.09) | 10.25 (3.86)
  Pre-treatment (IBS Group): number analyzed (Participants) | 6 | 2 | 5
  Pre-treatment (IBS Group) | 18.67 (11.08) | 17.00 (4.24) | 17.40 (7.30)
  Post-treatment (IBS Group): number analyzed (Participants) | 6 | 2 | 5
  Post-treatment (IBS Group) | 13.17 (7.41) | 16.00 (4.24) | 15.20 (10.18)

10. Secondary Outcome: Patient Assessment of Constipation - Quality of Life (PAC-QOL)
Description: Patient Assessment of Constipation Quality of Life Questionnaire. A validated questionnaire containing 28 total questions with four sub-sections each broadly ranging from "not at all" to "all of the time" on 0 to 4 scales.
  Possible total range is 0 to 112. An overall higher total score on the PAC-QOL means a worse outcome. PAC-QOL was completed at four time-points (Day -14, Day 0, Day 15, & Day 22). Scores were aggregated based on time period as either pre- (Day -14 & Day 0) or post- (Day 15 & Day 22) treatment start. Values reported are averages based on patient total scores from these time points. Data was specifically analyzed based on patient diagnosis in addition to treatment.
Time Frame: Day -14 to Day 22
Population: All participants who completed the study and had both pre and post treatment PAC-QOL ratings
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
score on a scale
  Pre-treatment (CIC Group): number analyzed (Participants) | 13 | 9 | 4
  Pre-treatment (CIC Group) | 39.08 (17.09) | 31.22 (6.57) | 26.50 (14.25)
  Post-treatment (CIC Group): number analyzed (Participants) | 13 | 9 | 4
  Post-treatment (CIC Group) | 26.46 (18.30) | 20.56 (4.42) | 19.75 (6.99)
  Pre-treatment (IBS Group): number analyzed (Participants) | 6 | 2 | 5
  Pre-treatment (IBS Group) | 41.00 (17.01) | 32.00 (4.24) | 34.30 (14.48)
  Post-treatment (IBS Group): number analyzed (Participants) | 6 | 2 | 5
  Post-treatment (IBS Group) | 30.33 (20.20) | 23.00 (1.41) | 35.60 (8.53)

11. Secondary Outcome: Need for Rescue Laxatives
Description: Number of total days that rescue laxatives were used by participants in each treatment group.
  (The number of days that rescue laxatives were used by each individual patient was calculated and added to the treatment group total)
Time Frame: 55 days (baseline, treatment, & follow-up)
Population: All participants who completed the study and had daily medication usage data
Measure: Number; unit: days
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
days | 13 | 6 | 3

12. Secondary Outcome: Spontaneous Bowel Movement (SBM) Frequency
Description: Average number of Spontaneous Bowel Movements per day. (Spontaneous Bowel Movements include both complete and incomplete bowel movements)
Time Frame: 55 days (baseline, treatment, & follow-up)
Population: All participants who completed the study and had both pre and post treatment SBM measurements
Measure: Mean (Standard Deviation); unit: number of SBMs per day
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
Number analyzed (Participants) | 19 | 11 | 9
number of SBMs per day
  Pre-treatment | 0.75 (0.29) | 0.70 (0.40) | 0.75 (0.39)
  Post-treatment | 0.95 (0.36) | 0.79 (0.35) | 0.89 (0.58)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each subject throughout the study duration, from study enrollment to final day in study (includes 9-day follow-up period). Study duration was approximately 46-59 days.
Description: All participants of the study were assessed for adverse events throughout the duration of the study. Adverse events were recorded, logged, and reported to the IRB where applicable. In-person follow-up was arranged for participants experiencing an adverse event to monitor resolution of symptoms.
Arm/Group | CSP01 | Carboxymethylcellulose (CMC) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 1/20 | 0/11 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSP01 (N=20) | Carboxymethylcellulose (CMC) (N=11) | Placebo (N=9)
Constipation and back pain caused by constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Subject experienced several bowel movements per day coupled with a sense of urgency, but never able to have a complete bowel movement. Subject also developed back pain attributed to constipation.

LIMITATIONS AND CAVEATS:
Target number of participants needed to achieve target power was not attained. One subject's post-treatment SmartPill data was irretrievable due to unexpected technical malfunction, therefore post-treatment colonic transit time was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT03054506/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT03054506/ICF_001.pdf